CLINICAL TRIAL: NCT06782178
Title: Temporomandibular Joint Arthroscopic Lysis and Lavage Compared to Arthrocentesis in Disc Displacement Without Reduction: a Randomised, Double-blind, Controlled Trial
Brief Title: TMJ Arthroscopy Compared to Arthrocentesis in Disc Displacement Without Reduction
Acronym: ACALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Eastmaninstitutet (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mattias Ulmner, Lecturer, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-06294-01
Record Dates: First submitted 2025-01-02; First posted 2025-01-17 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-01

CONDITIONS: Temporomandibular Joint Disc Displacement; Temporomandibular Joint Disc Displacement, Without Reduction; Temporomandibular Disorders (TMD)
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Therapeutic Irrigation; Arthrocentesis; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic lysis and lavage (Experimental)
  Interventions: Procedure: Arthroscopic lysis and lavage
- Arthrocentesis (Active Comparator)
  Interventions: Procedure: Arthrocentesis/Saline

INTERVENTIONS:
Procedure: Arthroscopic lysis and lavage — Arthroscopic lysis and lavage refers to an arthroscopic procedure where the temporomandibular joint is rinsed with saline solution and where the joint capsule is distended and where adhesions are lysated bluntly.
  Arms: Arthroscopic lysis and lavage
Procedure: Arthrocentesis/Saline — Arthrocentesis refers to a blind irrigation of the temproromandibular joint with saline solution
  Arms: Arthrocentesis

SUMMARY:
The goal of this clinical trial is to compare the intervention arthroscopic lysis and lavage to the intervention arthrocentesis in treating disabling and painful temporomandibular joint disc displacement without reduction. The main questions it aims to answer are:

* Which surgical method that best improves mouth opening capacity, TMJ pain, and TMJ disability?
* If any pre- or peri-operative variable/-s could be identified as a predictor for surgical outcome? Researchers will compare arthroscopic lysis and lavage to arthrocentesis to see if arthroscopic lysis and lavage works better to treat temporomandibular joint disc displacement.

Participants will:

* Have one of the two interventions under general anesthesia, not knowing which intervention.
* Visit an external clinic for regular checkups at 1, 3, 6, 12, and 24 months after surgery.
* Answer three different quality of life surveys at the checkups.

DETAILED DESCRIPTION:
1. BACKGROUND The temporomandibular joint (TMJ) is a bilateral joint comprised of two cartilage covered bone surfaces that articulates against each other during mouth opening and closing. A dense cartilage disc is situated between the two joint surfaces.

   Disc displacement (DD) is characterised by an improper position of the TMJ disc relative to the articulating surfaces and affects up to 30% of the population. DD without reduction (DDwoR) is a sub-diagnosis of DD where the inaccurate disc position and associated inflammation hampers the TMJ movement and osteoarthritis successively develops. The affected patient suffers from reduced mouth opening capacity and pain when opening the mouth and during chewing, which leads to restrains in food intake, speech and social activities. A recent Swedish publication has shown that patients with TMJ disorders had more days of work disability (2-3 times longer) compared to a non-TMD cohort followed over a ten year period. The reliance on social security benefits in the group of patients that had TMJ surgery more than once were more accentuated compared to other TMJ disorder patients.

   The primary treatment for DDwoR is non-surgical, i.e., physiotherapy, pharmacological treatment and/or occlusal splint therapy. If non-surgical treatment fails, arthroscopic lysis and lavage (ALL) or arthrocentesis (AC) might be considered. ALL is performed with a rod-shaped lens inserted into the TMJ cavity enabling direct visualisation, The operative procedure involves manipulation of disc position, release of adhesions (lysis), and irrigation (lavage) of the joint with either saline solution or Ringer's solution. Generally the procedure is performed under general anaesthesia, but there are reports on ALL performed in local anaesthesia or conscious sedation. Success rates of 75-88 % is reported. In AC, two needles are inserted into the joint cavity to irrigate the TMJ. The method does not allow visualisation of the joint. AC is often performed together with opening and closing manoeuvres of the mandible to enable manipulation of the discs position. AC is reported to be executed under general anaesthesia, but also under local anaesthesia or conscious sedation. AC is most often reported to have a higher success rate compared to ALL, with figures ranging from 66-100 %. Although, the compared figures are taken from cohort studies with no control group. There are a few randomised and controlled studies comparing ALL to AC. Fridrich et al. performed a randomised study without blinding and also incorporates two different diagnoses, DDwoR and disc displacement with reduction (DDwR). The patient sample was small, 20 patients. Murakami et al. conducted a study including three interventions: non-surgical , ALL and AC. The study was not blinded and not randomised, and 25 patients were included in the ALL-group and 20 patients in the AC group. The patients had the diagnosis DDwoR. In a third study, a total of 63 patients were treated, 33 had arthroscopy and 29 had arthrocentesis. The study was not blinded and 8 of the included patients was diagnosed with DDwR and the remaining with DDwoR. All three studies showed a better outcome for patients treated with arthroscopy, even though the result was not significant in two of the studies. In a meta-analysis published 2015 both MIO and patient-assessed TMJ pain had significantly better outcome in arthroscopy.

   Synovial fluid from the TMJ has been used since the mid-90's mostly for analysing inflammatory markers. Proteomics is a relatively new technique for analysing protein profiles and has only been applied a couple of times in the field of TMJ pathology. Since the aetiology of DD is still not known, proteomics provides a comprehensive insight of the protein profile of TMJ disorders.

   There are very few RCT's comparing the outcome of ALL and AC in patients with DDwoR and to this date none with a blinding. The aim of this study is to evaluate outcome of ALL and AC in treating DDwoR in a double-blind fashion. Another aim is to investigate synovial fluid protein profile in TMJ DD and to see if patient-specific differences might be connected to surgical outcome, local inflammation, local pain, or level of degenerative changes.
2. HYPOTHESIS/RESEARCH QUESTIONS ALL has a superior outcome compared to AC treating patients with DDwoR. The outcome will be longitudinally evaluated by maximum mouth opening capacity, patient reported TMJ pain and TMJ disability, and Quality of life (QoL) questionnaires at pre-determined time-points during a 24-month postoperative period.

   The primary research question is which surgical method that best improves the above stated variables.

   A secondary question is if there is an identifiable protein profile regarding DDwoR.

   A tertiary question is if any pre- or peri-operative variable/-s could be identified as a predictor for outcome.

   A quaternary is the impact from DDwoR on QoL and the surgical outcomes impact on QoL.

   A last question is if none of the therapies are better than the other, do the recovery time after surgery differ between ALL and AC.
3. METHODS 3.1. Study design

Randomised, double-blind, controlled study where the outcome of ALL and AC on patients with DDwoR is compared.

3.2. Data source

All patients referred to the Department of Oral- and Maxillofacial Surgery, Karolinska University Hospital, Stockholm, with the diagnosis DDwoR and with a history of not responding to non-surgical treatment will be screened for inclusion.

3.3. Exposure/Intervention

Patients will be assigned to either ALL or AC. Both treatments will be performed under general anaesthesia. The randomisation will be made in blocks of two in a 1:1 ratio. A computer software provided by KTA (Karolinska Trial Alliance) will handle the randomisation process. At time of surgery, when the patient is under general anaesthesia and draped in sterile cloth, the patient will be allocated to either ALL or AC. In this manner the intervention or placebo treatment will be blinded to the patient but not to the surgeon. The person evaluating the outcome of surgery (the assessor) will not know which treatment the patient has undertaken. The two surgical procedures are described below.

ALL: The surgical procedure is performed according to the original description of the technique. Local During the operation the joint space is irrigated with a minimum of 300 mL saline solution. A pressure infuser (InfuseITTM) set at 175 mmHg will be used to standardise the irrigation pressure. At the start of joint irrigation, the first 50 mL outflow irrigation fluid will be collected in a sterile container for later proteomic analysis. At the end of surgery, the joint is flushed with 10 mL of Marcaine-Adrenaline (2.5 mg/mL). No other medication will be injected or otherwise introduced into the joint compartment. The incision is sutured with a single non-resorbable suture, and a wound dressing is put over the incision. The described intervention is standardized and takes no more than 30 minutes.

AC: Arthrocentesis of the TMJ was first described in 1991 and the same technique is used here with the exception that no corticosteroids are injected in the joint postoperatively. During the operation the joint space is irrigated with a minimum of 300 mL saline solution. A pressure infuser (InfuseITTM) set at 175 mmHg will be used to standardise the irrigation pressure. At the start of joint irrigation, the first 50 mL outflow irrigation fluid will be collected in a sterile container for later proteomic analysis. After finishing the mandibular manipulation and the joint irrigation, the joint is flushed with 10 mL of Marcaine-Adrenaline (2.5 mg/mL). No other medication will be injected or otherwise introduced into the joint compartment. Finally, a vertical preauricular skin incision (approximately 5 mm long) is made to mimic an arthroscopic procedure. The incision is sutured with a single non -resorbable suture and a wound dressing is put over the incision.

To keep the blinding intact for the patient and the assessor, the medical chart will be written as if all the patients had AC performed.

Both the intervention groups will have postoperative physiotherapy training for a period of one month from the day after surgery in accordance with a specified home exercise program (see attachment). If needed, the home exercise program can be prolonged or individually adjusted after the first month. If the patient uses an occlusal splint prior to surgery the splint may have to be adjusted and that has to be performed by the assessor.

3.4. Outcome

Please see "Outcome measure" below.

3.5. Sample size

50 patients in each intervention group, i.e., 100 patients in total, in accordance with the power analysis, see "Statistical analysis".

3.6. Inclusion and exclusion criteria

Please, see "Eligibility" below.

3.7. Data collection

At registration for surgery and after obtained informed consent, baseline data is collected by the surgeon designating the patient to surgery. Predetermined follow-up visits are at 1 week when the surgeon will remove the stich and do a reinstruction for the home-exercise program, and at 1, 3, 6, 12 and 24 months postoperative when the assessor examine the patient according to the specific exam protocol (see attachment) The assessor/-s will be calibrated alongside the surgeon/-s before the start of the study in accordance with the DC/TMD criteria. At 6-month intervals the surgeons and assessors will have a meeting for re-calibrating purposes.

Objective data only registered preoperative: name, personal identification number, age, sex, affected joint (left, right).

Objective data registered both pre- and post-operatively: MIO with and without pain (mm), lateral excursive movement (mm), protrusion (mm), pain upon palpating masticatory muscles, pain upon lateral joint palpation.

Subjective data registered both pre- and post-operatively: patient-reported TMJ disability (NRS 0-10), patient-reported TMJ pain (NRS 0-10), patient-reported psycho-social impairment because of TMJ disorder (NRS 0-10), patient-reported global pain (NRS 0-10), and quality of life questionnaire EQ-5D-5L, JFSL-8, and OHIP 14-S.

Perioperative data: antibiotic prophylaxis (yes/no), performed surgery (AC/ALL), maximum assisted mouth opening (mm), duration of surgery (min), duration of general anaesthesia (min), lavage volume (mL), preauricular swelling due to lavage (yes/no),Wilkes grading (3-5), negative event during and due to surgery. Grading of intraarticular conditions will be made according to the scale proposed by Gynther et al.: synovitis (0-3), degenerative changes (0-3), and fibrosis/adhesions (0-2), in case of ALL.

3.8. Revelation of blinding At the 6-month visit the patients will be asked if they believe that they had ALL or AC. The assessor will also give their opinion in that matter. After the 6-month follow-up, the blinding will be revealed to the patient if they want to. Patients with a non-successful outcome might be offered another therapy; non-surgical or surgical. Controls will be made at 12- and 24-months post-operative regarding all patients.

3.9. Analysis of synovial fluid Proteomic analysis and protein quantification in synovial fluid will be performed at PainOmics laboratory, University hospital in Linköping. In this project, we will follow a discover and verification/validation schema. In the first step peptides and protein contents of the synovial fluid will be analysed using 2-DE in combination with mass spectrometry. With this technique it is possible to separate and quantify more than 1000 proteins and it is the only technique that allows separating and studying different protein isoforms. Quantification of the separated proteins is achieved by spot integration using specialized 2-DE software that makes it possible to compare protein patterns from different subjects/groups. Identification of the protein is performed by in-gel digestion of each protein, recovery of the fragments from the gel, and analysis by mass spectrometry (MS) using MALDI-T

4. STATISTICAL ANALYSIS The primary objective is to evaluate the superiority of ALL compared to AC in patients diagnosed with DDwoR and not responding to non-surgical treatment. The outcome variable is dichotomous (successful/not successful) where a successful outcome in the ALL group is assessed to be 80 % and in the AC group 50 %. With 80 % power and a 5 % significance level the groups must contain 45 patients each. Dropout rate of 10 % is accounted for which means that 50 patients/group must be included to verify superiority.

Statistical analyses will be performed using the Chi-Square test for bivariate data and the Students t-test (unpaired and paired) for mean values, as well as repeated measures ANOVA. Longitudinal data will be analysed with linear regression analysis and predictors for surgical outcome will be evaluated through logistic regression. The intention to treat analysis model will be used.

Potential known confounders may be adjusted for in the analysis and the risk of residual unknown confounders should be reduced by the randomisation process.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral DDwoR affecting the patients mouth opening capacity to a range of ≤ 35 mm, verified with clinical and magnetic resonance imaging (MRI) findings.
* TMJ pain ≥ 3 (NRS)
* TMJ disability ≥ 3 (NRS)
* Age ≥ 18 years

Exclusion Criteria:

* Prior open TMJ surgery
* Patient diagnosed with rheumatologic joint disease.
* ASA (American Society of Anaesthesiologists) > 3
* Patient unable to verify informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Treatment outcome | From intervention to the 6 month postoperative follow up.
  The three criteria below have to be fulfilled to verify a good treatment outcome.
  1. Maximum interincisal opening (MIO) of ≥ 35 mm, or an increase of MIO of ≥ 40 %.
  2. Patient-reported TMJ pain. Visual analogue scale (VAS) ≤ 3, or ≤ 40% reduction.
  3. Patient-reported TMJ disability. VAS ≤ 3, or a 40 % reduction.

SECONDARY OUTCOMES:
Qulity of life surveys | From intervention to the 6 month postoperative follow up.
  to evaluate EQ-5D-5L, JFSL-8, and OHIP 14-S and what impact DDwoR has got on QoL and difference in QoL after intervention.

OTHER OUTCOMES:
Pain in the temporomandibular joint (TMJ) during function | From intervention to the 6 month postoperative follow up.
  The patient is asked to estimate how much pain TMJ function (opening, biting, chewing, speaking, etc.) has caused on average over the past 2-week period. This estimation should exclude the worst imaginable pain. Each TMJ is assessed individually, meaning the patient should provide a numerical value between 0 (no pain) and 10 (worst imaginable pain) for each joint.
Pain in the temporomandibular joint at rest | From intervention to the 6 month postoperative follow up.
  The patient is asked to estimate pain in each TMJ at rest on a scale graded from 0 to 10. The value should reflect an average representative of the past 2-week period.
Functional impairment of the temporomandibular joint | From intervention to the 6 month postoperative follow up.
  The patient is asked to estimate the degree of functional impairment caused by current TMJ issues. This variable includes both joint mobility and the ability to consume food. The scale is graded from 0 to 10. A score of 0 indicates no impairment, meaning unrestricted jaw opening and the ability to eat all types of food without difficulty. A score of 10 represents complete functional impairment, such as zero millimeters of opening or being able to consume only liquids due to the inability to chew solid food.
Psychosocial impact | From intervention to the 6 month postoperative follow up.
  The patient is asked to estimate the psychosocial impact of their TMJ issues from 0 to 10. A score of 0 indicates no impact, while a score of 10 represents the worst imaginable impact. This may include how much and how often the patient thinks about their TMJ issues, how it affects their mood, and how it impacts their social life, such as withdrawing from social interactions.
Other bodily pain | From intervention to the 6 month postoperative follow up.
  The patient is asked to estimate the degree of bodily pain unrelated to TMJ pain between 0 to 10. This can include pain from other joints, gastrointestinal discomfort, etc. A score of 0 indicates no other bodily pain, while a score of 10 indicates the worst imaginable bodily pain.
Palpation tenderness of TMJ | From intervention to the 6 month postoperative follow up.
  The TMJ is palpated laterally according to DC/TMD (500 grams pressure). A letter balance is used to calibrate palpation pressure. The pain must be recognizable to the patient.
Palpation tenderness of the masseter and temporalis muscles | From intervention to the 6 month postoperative follow up.
  The masseter and temporalis muscles are palpated at three separate sites each, according to DC/TMD (1000 grams pressure). A letter balance is used to calibrate palpation pressure. The pain must be recognizable to the patient.
Maximum interincisal opening (MIO) | From intervention to the 6 month postoperative follow up.
  Measured in millimeters. The distance between teeth 11 and 41 is measured as the patient opens their mouth as wide as possible. If this is not feasible due to malocclusion, tooth loss, etc., an alternative representative pair of front teeth is chosen for measurement. This should be noted in the patient's record to ensure consistent measurements in the future.
Maximum protrusion | From intervention to the 6 month postoperative follow up.
  Horizontal overbite (HOB) is first measured in millimeters during habitual intercuspal position. The value is positive if tooth 11 is located facially to tooth 41 and negative if the reverse is true. The patient is then instructed to protrude the mandible maximally, and the horizontal distance between the incisal edges of teeth 11 and 41 is measured again. These two measurements are then added together (noting negative HOB in Class III cases).
Maximum laterotrusion | From intervention to the 6 month postoperative follow up.
  The patient is instructed to move the mandible to one side. The distance between the midline of the maxilla (between teeth 11 and 21) and the midline of the mandible (between teeth 31 and 41) is measured in millimeters. Any midline deviation during habitual intercuspal position is measured and subtracted from or added to the recorded value. Laterotrusion is measured for both left and right movements.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Ulmner, DDS, PhD, Principal Investigator — Karolinska Institutet, Department of Dental Medicine
Locations (1):
- Karolinska Institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and SAP is available through ClinicalTrials.

REFERENCES:
- [Background] Wilkes CH. Internal derangements of the temporomandibular joint. Pathological variations. Arch Otolaryngol Head Neck Surg. 1989 Apr;115(4):469-77. doi: 10.1001/archotol.1989.01860280067019. PMID 2923691
- [Background] Ulmner M, Weiner CK, Lund B. Predictive factors in temporomandibular joint arthroscopy: a prospective cohort short-term outcome study. Int J Oral Maxillofac Surg. 2020 May;49(5):614-620. doi: 10.1016/j.ijom.2019.09.002. Epub 2019 Sep 26. PMID 31564479
- [Background] Ulmner M, Sugars R, Naimi-Akbar A, Alstergren P, Lund B. Cytokines in temporomandibular joint synovial fluid and tissue in relation to inflammation. J Oral Rehabil. 2022 Jun;49(6):599-607. doi: 10.1111/joor.13321. Epub 2022 Apr 9. PMID 35342975
- [Background] Ulmner M, Kruger-Weiner C, Lund B. Patient-Specific Factors Predicting Outcome of Temporomandibular Joint Arthroscopy: A 6-Year Retrospective Study. J Oral Maxillofac Surg. 2017 Aug;75(8):1643.e1-1643.e7. doi: 10.1016/j.joms.2017.04.005. Epub 2017 Apr 13. PMID 28487216
- [Background] Tuz HH, Baslarli O, Adiloglu S, Gokturk T, Meral SE. Comparison of local and general anaesthesia for arthrocentesis of the temporomandibular joint. Br J Oral Maxillofac Surg. 2016 Oct;54(8):946-949. doi: 10.1016/j.bjoms.2016.06.026. Epub 2016 Jul 18. PMID 27435500
- [Background] Smolka W, Yanai C, Smolka K, Iizuka T. Efficiency of arthroscopic lysis and lavage for internal derangement of the temporomandibular joint correlated with Wilkes classification. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Sep;106(3):317-23. doi: 10.1016/j.tripleo.2007.12.007. Epub 2008 Jan 15. PMID 18226569
- [Background] Sanders B. Arthroscopic surgery of the temporomandibular joint: treatment of internal derangement with persistent closed lock. Oral Surg Oral Med Oral Pathol. 1986 Oct;62(4):361-72. doi: 10.1016/0030-4220(86)90282-3. PMID 3464910
- [Background] Salinas Fredricson A, Kruger Weiner C, Adami J, Rosen A, Lund B, Hedenberg-Magnusson B, Fredriksson L, Svedberg P, Naimi-Akbar A. Sick leave and disability pension in a cohort of TMD-patients - The Swedish National Registry Studies for Surgically Treated TMD (SWEREG-TMD). BMC Public Health. 2022 May 9;22(1):916. doi: 10.1186/s12889-022-13329-z. PMID 35534826
- [Background] Sale H, Bryndahl F, Isberg A. Temporomandibular joints in asymptomatic and symptomatic nonpatient volunteers: a prospective 15-year follow-up clinical and MR imaging study. Radiology. 2013 Apr;267(1):183-94. doi: 10.1148/radiol.12112243. Epub 2012 Dec 18. PMID 23249569
- [Background] Olsen-Bergem H, Bjornland T. A cohort study of patients with juvenile idiopathic arthritis and arthritis of the temporomandibular joint: outcome of arthrocentesis with and without the use of steroids. Int J Oral Maxillofac Surg. 2014 Aug;43(8):990-5. doi: 10.1016/j.ijom.2014.03.018. Epub 2014 May 1. PMID 24794763
- [Background] Nogueira EFC, Lemos CAA, Vasconcellos RJH, Moraes SLD, Vasconcelos BCE, Pellizzer EP. Does arthroscopy cause more complications than arthrocentesis in patients with internal temporomandibular joint disorders? Systematic review and meta-analysis. Br J Oral Maxillofac Surg. 2021 Dec;59(10):1166-1173. doi: 10.1016/j.bjoms.2021.05.007. Epub 2021 May 15. PMID 34274169
- [Background] Nitzan DW, Samson B, Better H. Long-term outcome of arthrocentesis for sudden-onset, persistent, severe closed lock of the temporomandibular joint. J Oral Maxillofac Surg. 1997 Feb;55(2):151-7; discussion 157-8. doi: 10.1016/s0278-2391(97)90233-0. PMID 9024352
- [Background] Nitzan DW, Dolwick MF, Martinez GA. Temporomandibular joint arthrocentesis: a simplified treatment for severe, limited mouth opening. J Oral Maxillofac Surg. 1991 Nov;49(11):1163-7; discussion 1168-70. doi: 10.1016/0278-2391(91)90409-f. PMID 1941330
- [Background] Murakami K, Hosaka H, Moriya Y, Segami N, Iizuka T. Short-term treatment outcome study for the management of temporomandibular joint closed lock. A comparison of arthrocentesis to nonsurgical therapy and arthroscopic lysis and lavage. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1995 Sep;80(3):253-7. doi: 10.1016/s1079-2104(05)80379-8. PMID 7489265
- [Background] Mehra P, Arya V. Temporomandibular joint arthrocentesis: outcomes under intravenous sedation versus general anesthesia. J Oral Maxillofac Surg. 2015 May;73(5):834-42. doi: 10.1016/j.joms.2014.11.018. Epub 2014 Dec 31. PMID 25795184
- [Background] Machon V, Sedy J, Klima K, Hirjak D, Foltan R. Arthroscopic lysis and lavage in patients with temporomandibular anterior disc displacement without reduction. Int J Oral Maxillofac Surg. 2012 Jan;41(1):109-13. doi: 10.1016/j.ijom.2011.07.907. Epub 2011 Sep 1. PMID 21885248
- [Background] Liu X, Yang Y, Chen L, Tian S, Abdelrehem A, Feng J, Fu G, Chen W, Ding C, Luo Y, Zou D, Yang C. Proteome Analysis of Temporomandibular Joint with Disc Displacement. J Dent Res. 2022 Dec;101(13):1580-1589. doi: 10.1177/00220345221110099. Epub 2022 Oct 20. PMID 36267015
- [Background] Kellesarian SV, Al-Kheraif AA, Vohra F, Ghanem A, Malmstrom H, Romanos GE, Javed F. Cytokine profile in the synovial fluid of patients with temporomandibular joint disorders: A systematic review. Cytokine. 2016 Jan;77:98-106. doi: 10.1016/j.cyto.2015.11.005. Epub 2015 Nov 7. PMID 26556103
- [Background] Kaneyama K, Segami N, Sun W, Sato J, Fujimura K. Analysis of tumor necrosis factor-alpha, interleukin-6, interleukin-1beta, soluble tumor necrosis factor receptors I and II, interleukin-6 soluble receptor, interleukin-1 soluble receptor type II, interleukin-1 receptor antagonist, and protein in the synovial fluid of patients with temporomandibular joint disorders. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Mar;99(3):276-84. doi: 10.1016/j.tripleo.2004.06.074. PMID 15716832
- [Background] Jasim H, Ernberg M, Carlsson A, Gerdle B, Ghafouri B. Protein Signature in Saliva of Temporomandibular Disorders Myalgia. Int J Mol Sci. 2020 Apr 7;21(7):2569. doi: 10.3390/ijms21072569. PMID 32272779
- [Background] Holmlund A, Gynther G, Axelsson S. Efficacy of arthroscopic lysis and lavage in patients with chronic locking of the temporomandibular joint. Int J Oral Maxillofac Surg. 1994 Oct;23(5):262-5. doi: 10.1016/s0901-5027(05)80104-3. PMID 7890964
- [Background] Herr MM, Fries KM, Upton LG, Edsberg LE. Potential biomarkers of temporomandibular joint disorders. J Oral Maxillofac Surg. 2011 Jan;69(1):41-7. doi: 10.1016/j.joms.2010.05.013. PMID 21163381
- [Background] Gynther GW, Holmlund AB, Reinholt FP, Lindblad S. Temporomandibular joint involvement in generalized osteoarthritis and rheumatoid arthritis: a clinical, arthroscopic, histologic, and immunohistochemical study. Int J Oral Maxillofac Surg. 1997 Feb;26(1):10-6. doi: 10.1016/s0901-5027(97)80838-7. PMID 9081245
- [Background] Gynther GW, Holmlund AB, Reinholt FP. Synovitis in internal derangement of the temporomandibular joint: correlation between arthroscopic and histologic findings. J Oral Maxillofac Surg. 1994 Sep;52(9):913-7; discussion 918. doi: 10.1016/s0278-2391(10)80066-7. PMID 8064453
- [Background] Grossmann E, Poluha RL, Iwaki LCV, Santana RG, Iwaki Filho L. The use of arthrocentesis in patients with temporomandibular joint disc displacement without reduction. PLoS One. 2019 Feb 13;14(2):e0212307. doi: 10.1371/journal.pone.0212307. eCollection 2019. PMID 30759144
- [Background] Goudot P, Jaquinet AR, Hugonnet S, Haefliger W, Richter M. Improvement of pain and function after arthroscopy and arthrocentesis of the temporomandibular joint: a comparative study. J Craniomaxillofac Surg. 2000 Feb;28(1):39-43. doi: 10.1054/jcms.1999.0103. PMID 10851672
- [Background] Fu K, Ma X, Zhang Z, Chen W. Tumor necrosis factor in synovial fluid of patients with temporomandibular disorders. J Oral Maxillofac Surg. 1995 Apr;53(4):424-6. doi: 10.1016/0278-2391(95)90717-3. PMID 7699497
- [Background] Fridrich KL, Wise JM, Zeitler DL. Prospective comparison of arthroscopy and arthrocentesis for temporomandibular joint disorders. J Oral Maxillofac Surg. 1996 Jul;54(7):816-20; discussion 821. doi: 10.1016/s0278-2391(96)90526-1. PMID 8676225
- [Background] Emshoff R, Rudisch A. Temporomandibular joint internal derangement and osteoarthrosis: are effusion and bone marrow edema prognostic indicators for arthrocentesis and hydraulic distention? J Oral Maxillofac Surg. 2007 Jan;65(1):66-73. doi: 10.1016/j.joms.2005.11.113. PMID 17174766
- [Background] Doetzer AD, Herai RH, Buzalaf MAR, Trevilatto PC. Proteomic Expression Profile in Human Temporomandibular Joint Dysfunction. Diagnostics (Basel). 2021 Mar 28;11(4):601. doi: 10.3390/diagnostics11040601. PMID 33800589
- [Background] Carvajal WA, Laskin DM. Long-term evaluation of arthrocentesis for the treatment of internal derangements of the temporomandibular joint. J Oral Maxillofac Surg. 2000 Aug;58(8):852-5; discussion 856-7. doi: 10.1053/joms.2000.8201. PMID 10935583
- [Background] Briggs KA, Breik O, Ito K, Goss AN. Arthrocentesis in the management of internal derangement of the temporomandibular joint. Aust Dent J. 2019 Mar;64(1):90-95. doi: 10.1111/adj.12665. Epub 2018 Dec 19. PMID 30422323
- [Background] Breik O, Devrukhkar V, Dimitroulis G. Temporomandibular joint (TMJ) arthroscopic lysis and lavage: Outcomes and rate of progression to open surgery. J Craniomaxillofac Surg. 2016 Dec;44(12):1988-1995. doi: 10.1016/j.jcms.2016.09.017. Epub 2016 Oct 5. PMID 27836550
- [Background] Al-Moraissi EA, Wolford LM, Ellis E 3rd, Neff A. The hierarchy of different treatments for arthrogenous temporomandibular disorders: A network meta-analysis of randomized clinical trials. J Craniomaxillofac Surg. 2020 Jan;48(1):9-23. doi: 10.1016/j.jcms.2019.10.004. Epub 2019 Nov 5. PMID 31870713
- [Background] Abboud WA, Givol N, Yahalom R. Arthroscopic lysis and lavage for internal derangement of the temporomandibular joint. Ann Maxillofac Surg. 2015 Jul-Dec;5(2):158-62. doi: 10.4103/2231-0746.175754. PMID 26981463
- [Background] Al-Moraissi EA. Arthroscopy versus arthrocentesis in the management of internal derangement of the temporomandibular joint: a systematic review and meta-analysis. Int J Oral Maxillofac Surg. 2015 Jan;44(1):104-12. doi: 10.1016/j.ijom.2014.07.008. Epub 2014 Aug 7. PMID 25123511